CLINICAL TRIAL: NCT04011917
Title: Projected Prognosis as a Predictor of Short-term Outcome After Treatment of Minor Musculoskeletal Injuries in the Emergency Department: A Prospective Cohort Study
Brief Title: Projected Prognosis as a Predictor of Short-term Outcome After Treatment of Minor Musculoskeletal Injuries in the Emergency Department
Status: Completed | Type: Observational
Sponsor: Slagelse Hospital (Other)
Collaborators: Bispebjerg Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: REG-032-2019
Record Dates: First submitted 2019-07-04; First posted 2019-07-09 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Musculoskeletal Diseases
Keywords: Minor Musculoskeletal Injuries; Emergency Department; Prediction outcome; Extended Scope Physiotherapists
MeSH Terms: conditions — Musculoskeletal Diseases; Emergencies | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Caseload group
  Interventions: Behavioral: Standard care
- Prediction group
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Behavioral: Standard care — Treatment by an extended scope physiotherapist following Standard Operating Procedures.

SUMMARY:
This study describes the caseload treated by the extended scope physiotherapists(ESP) working in the emergency department at Slagelse Hospital.

Patients treated by the ESP during a 3 month period will be included in this study.

Furthermore we aim to assess if ESPs treating patients with minor musculoskeletal injuries in the ED can predict the short-term prognosis of recovery. The prediction is made at hospital discharge using a (-7/+7) numerical rating scale (-7=poor prognosis; 7=best prognosis).

ELIGIBILITY:
Inclusion Criteria:

* 1 Treated by an ESP for a minor musculoskeletal injury in the emergency room
* 2 Has an email address
* 3 Signed informed consent form

Exclusion Criteria:

* 1 A condition that, in the opinion of the investigator, would preclude participation in the study (e.g., not having access to the internet, cognitive impairments etc.)
* 2 Under the influence of drugs or alcohol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients treated by an ESP physiotherapist in the emergency room at Slagelse Hospital, Denmark, in a 3 month period +1 month follow-up will be invited to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 432 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Transition ratings of global perceived effect | 1 month after discharge
  Using a transition questionnaire (TRANS-Q) the perceived effect of treatment will be measured by participants answering if their current health status is "unchanged", "worse" or "better" compared to their pre-injury status. "unchanged" equals a transition score of 0. If the participant answers "worse", he/she is asked to rate the degree of worsening on a 7 point Likert scale, with corresponding scores ranging from -1 to -7. If the participant answers "better", he/she is asked to rate the degree of improvement on a 7 point Likert scale, with corresponding scores ranging from 1 to 7. Thus the GPE score range from -7 (worsening) to 7 (improvement), with the mid-point - 0 - representing no change.

SECONDARY OUTCOMES:
Patient Acceptable Symptom State | 1 month after discharge
EuroQoL questionnaire | 1 month after discharge

OTHER OUTCOMES:
VAS Pain | At baseline and 1 month after discharge
  The VAS pain is a measure of pain intensity, which has been widely used in diverse adult populations. The scale is a unidimensional continuous scale comprised of a horizontal line, anchored by 2 verbal descriptors, one for each symptom extreme (0 no pain, 10 the worst imaginable pain).
Analgesic use | 1 month after discharge
  The participants self-reported use of analgesics will be collected at the 1 month follow-up. Participants will be asked to note their use of analgesic drugs, within the week before the follow-up, only related to the treated injury in the emergency room.
Follow-up treatments | 1 month after discharge
  The participants self-reported use of follow-up visits with other allied health professionals will be recorded. All visits related to the treated injury during the 1-month follow-up period should be noted.
Re-injury | 1 month after discharge
  The participants self-reported reinjury rate during the 1-month follow-up period will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Christian P Olsen, PT, Phd candidate, Principal Investigator — Næstved-Slagelse-Ringsted Hospitals; Marius Henriksen, PT, PhD, Study Chair — Department of Physical and Occupational Therapy, Bispebjerg-Frederiksberg Hospital; Søren T Skou, PT, PhD, Study Chair — Næstved-Slagelse-Ringsted Hospitals and University of Southern Denmark
Locations (1):
- The Emergency Department, Slagelse Hospital, Slagelse, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Upon finalisation of the prespecified analyses we will share the IPD to other researchers based on an email inquiry.